CLINICAL TRIAL: NCT06944964
Title: Single vs. Dual Implant Fixation for Distal Femur Fractures in Older or Compromised Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFF Feasibility Study
Record Dates: First submitted 2025-03-04; First posted 2025-04-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Distal Femur Fractures
Keywords: Single Implant Fixation; Dual Implant Fixation; Dual Plate Fixation; Combination nail-plate fixation
MeSH Terms: conditions — Femoral Fractures, Distal

STUDY DESIGN:
Intervention Model Description: A multi-centered, preliminary feasibility RCT across 4 level I trauma centers comparing SIF to DIF for DFFs. Participants are randomized into one of two groups, and each group receives a different intervention (Single Implant Fixation (SIF) or Dual Implant Fixation (DIF)).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Control): Single Implant Fixation (SIF) (Active Comparator): Patients in this arm will undergo fixation of distal femur fractures using a single implant, which could be a lateral locked plate or a retrograde intramedullary nail.
  Interventions: Procedure: Single Implant Fixation (SIF)
- Group B (Experimental): Dual Implant Fixation (DIF) (Active Comparator): Patients in this arm will undergo fixation using dual implants, either dual plate fixation or a combination of nail and plate fixation.
  Interventions: Procedure: Dual Implant Fixation (DIF)

INTERVENTIONS:
Procedure: Single Implant Fixation (SIF) — This intervention involves using one implant for fracture fixation. The implant can be either a lateral locked plate or a retrograde intramedullary nail, based on the surgeon's preference.
  Arms: Group A (Control): Single Implant Fixation (SIF)
Procedure: Dual Implant Fixation (DIF) — This intervention involves using two implants for fracture fixation. The combination can be either dual plate fixation (DPF) or combination nail plate fixation (NPF) .
  Arms: Group B (Experimental): Dual Implant Fixation (DIF)

SUMMARY:
The goal of this clinical trial is to assess the feasibility of conducting a larger study comparing single implant fixation (SIF) and dual implant fixation (DIF) for treating distal femur fractures (DFF) in older or compromised adults. It will also evaluate the safety and effectiveness of these treatments. The main questions it aims to answer are:

* Can DIF improve patient outcomes compared to SIF in older or compromised adults?
* How feasible is it to recruit and retain participants for this trial?

Participants will:

1. Be randomly assigned to receive either SIF or DIF for their DFF treatment
2. Visit the clinic for follow-ups and assessments of their recovery and bone healing, including potential ultrasound imaging for detecting complications like non-union.

DETAILED DESCRIPTION:
The Investigators aim to conduct a multi-centre, preliminary RCT to determine the feasibility and inform the design of a definitive trial comparing patient-important outcomes between patients aged 40 years and older with distal femur fractures managed with SIF vs. DIF.

Primary Aim: Evaluate the feasibility of conducting a larger, definitive trial examining outcomes following SIF vs. DIF for DFFs in older or compromised adults. Our primary outcomes for this objective will be 1) recruitment and retention at the participating sites; and 2) site investigator feedback regarding barriers to protocol adherence.

Secondary Aims: Pilot the collection of candidate outcome measures to determine the optimal primary end point and sample size for a definitive trial. Our primary outcome for this objective will be the Oxford Knee Score, and secondary outcomes will include a range of patient-reported quality of life (QOL) measures, and objective clinical measures.

In addition, the study includes an ultrasound sub-study aimed at evaluating the feasibility of using ultrasound imaging to monitor bone healing and detect complications like non-union in patients with DFF.

Participants will be randomly assigned to receive either SIF or DIF, with SIF generally involving a single implant (such as a lateral locked plate or retrograde intramedullary nail) and DIF using a combination of implants (e.g., dual plates or a nail and plate). This randomized design will enable us to assess whether dual implant fixation offers improved clinical outcomes, such as reduced morbidity and faster weight-bearing recovery, compared to the more traditional single implant fixation.

Non-Randomized Participation: The investigators will collect data surrounding the number of eligible patients approached for consent, eligible patients not approached for consent and reason why, along with the proportion of patients who do not consent and reasons why to refine our strategy for the definitive trial. For patients who are excluded due to a lack of clinical equipoise, the investigators will provide the option of participating in a concurrent cohort study.This study will record the same variables as the RCT.

The trial will take place at four major trauma centers across Canada: London Health Sciences Centre - Victoria Hospital, St. Michael's Hospital, Sunnybrook Health Sciences Centre, and Alberta Health Services Centre. Participants will receive follow-up visits at these centers, which will include clinical check-ups, rehabilitation sessions, and imaging assessments to track their recovery progress.

The data gathered from this feasibility study will provide critical insights into the practicality of a larger-scale trial and will help inform future treatment strategies for distal femur fractures.

ELIGIBILITY:
Inclusion Criteria:

1. Isolated DFF (native AO/OTA-type A2, A3, C or periprosthetic Lewis and

   Rorabeck type 1, 2) and either:
   1. Age ≥ 60 years or;
   2. Age 18-60 years with one or more of:

   i. Osteoporosis ii. Obesity (Body Mass Index >30) iii. Metaphyseal comminution iv. Diabetes
2. Fracture amenable to plating and nailing
3. Ability to read and speak English or availability of a translator
4. Acute fractures (within 14-days of injury)
5. No surgeon preference regarding SIF vs. DIF
6. Provision of informed consent

Exclusion Criteria:

1. Candidate for primary or revision arthroplasty (surgeon opinion)
2. Periprosthetic fracture with loose implant
3. Gustillo grade III open fractures
4. Ipsilateral hip implant
5. Likely problems, in the judgment of the investigators, with maintaining follow-up (i.e., no fixed address, mentally competent to give consent, etc.)
6. Non-ambulatory patients
7. Multi-trauma patient (Injury Severity Score ≥ 16)
8. Lack of bone substance or poor bone-quality which, in the surgeon's judgment, makes fixation impossible
9. Any concomitant lower-extremity injury
10. Inability to obtain informed consent due to language barrier

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility Outcomes - Recruitment | Through study completion, an average of 1 year.
  Recruitment - 1) Recruitment (number of patients enrolled per-month). Success will be considered as each site enrolling a minimum mean of 0.6 patients per-month. This is a conservative estimate based on our previous trials in similar populations, and we expect that each site will screen a minimum of twice this number.
  * Number of patients enrolled per month
  * Success if each site able to enroll mean of 0.6 patients per month
Feasibility Outcomes - Retention | Through study completion, an average of 1 year.
  Retention - (proportion of patients that complete one-year follow-up). Success will be considered a minimum of 85% of patients with complete one-year data.
  * Proportion of patients that complete 1 year follow up
  * Success: 85%
Functional Ability | 2 year
  Via the validated Oxford Knee Score. It ranges from 0 to 48, with higher scores indicating better outcomes (i.e., less pain and better function).

SECONDARY OUTCOMES:
Pain rating | 2 years
  Via the numeric pain rating scale (NRS). 0-10; higher scores = worse pain.
Functional ability | 2 years
  Via the PROMIS-Physical Function Short. Higher = better for function domains
  Higher = worse for symptom domains (e.g., pain, fatigue).
  Form.
Weight-bearing | 2 years
  Using the Function IndeX for Trauma (FIX-IT) score.0-100; higher scores = better function.
Mobility | 3, 6, 12 and 24 months.
  Via the Extended Timed Up and Go (TUG) test starting at 3-months.
Health-related quality of life (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). | 2 years
  via Euro-Qol 5 Dimension (EQ5D). Higher scores = better health-related quality of life.
Health-resource utilization | 2 years
  Using the patient-reported Ambulatory and Home Care Record.
Complications | 2 years
  Including non-union, malunion, infection, implant failure and arthritis.
Re-operations (Type) | 2 years
  Reviewing the type of secondary procedure
Re-operations (Reason) | 2 years
  Reviewing the reason for the secondary procedure
Radiographic | 2 years
  To assess fracture healing and union. Anteroposterior and lateral x-rays of all patients will be obtained at the standard follow-up intervals. The independent adjudication committee will assess fracture healing and union.
Successful initiation of sites | Through study completion, an average of 24 months.
  Site fully approved, trained, and ready to begin recruiting participants.
Data quality | Through study completion, an average of 24 months.
  Proportion of CRFs with no missing data/outstanding queries
Randomization errors/cross-overs | Through study completion, an average of 24 months.
  Success: <5%, at least 90% adherence to allocated surgical technique
The proportion of patients instructed to WBAT in each group | Through study completion, an average of 24 months.
  Success: a minimum of 80% of patients are instructed to WBAT postoperative in each group
Barriers to protocol adherence | Through study completion, an average of 24 months.
  qualitative

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Fraser Orthopaedic Institute, New Westminster, British Columbia
  - London Health Sciences Centre, London, Ontario

IPD SHARING:
Plan to Share IPD: No